CLINICAL TRIAL: NCT02285881
Title: Shared Decision Making in Type 2 Diabetes With a Support Decision Tool That Takes Into Account Patient Preferences, Clinical Factors and the Intensity of Treatment: Design of a Cluster Randomised Trial
Brief Title: Shared Decision Making Between Patients and GPs in the Treatment of Type 2 Diabetes in Primary Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Rimke Vos, PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL39039.041.11
Record Dates: First submitted 2014-09-05; First posted 2014-11-07 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes treatment; personalized medicine; shared decision making; goal setting
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- shared decision making (Experimental): In the intervention practices the SDM process is used. In the SDM proces the patient and GP use a decision aid to discuss the pros and cons of two evidence based treatment possibilities, according to the Dutch College of General Practitioners (NHG) versus the ADDITION guideline, and the patients' preferences for either of these treatments. Together they choose one of these treatments, and set the five treatment targets (blood pressure, cholesterol, HbA1c, smoking status and weight) in order of priority. Subsequent treatment will take place according to the priorities of these OPTIMAL treatment targets. The priorities will be evaluated every 12 months.
  Interventions: Behavioral: Shared decision making
- control group (No Intervention): Patients in the control practices will receive treatment-as-before, which means that the patients will not be offered the structured SDM process. So the GP will treat the former ADDITION patients as they were used during the period that followed after the ADDITION study (2009), either according to the national guidelines or to the ADDITION intensive treatment algorithm.

INTERVENTIONS:
Behavioral: Shared decision making — In the intervention practices the SDM process is used. In the SDM proces the patient and GP use a decision aid to discuss the pros and cons of two evidence based treatment possibilities, according to the Dutch College of General Practitioners (NHG) versus the ADDITION guideline, and the patients' preferences for either of these treatments. Together they choose one of these treatments, and set the five treatment targets (blood pressure, cholesterol, HbA1c, smoking status and weight) in order of priority. Subsequent treatment will take place according to the priorities of these OPTIMAL treatment targets. The priorities will be evaluated every 12 months.
  Arms: shared decision making

SUMMARY:
Background: Less than 20% of type 2 diabetes mellitus (T2DM) patients in different healthcare settings achieve all treatment goals to prevent cardiometabolic disease. A more personalised approach with shared decision making should increase that percentage. Because the ADDITION-Europe study demonstrated two (almost) equally effective treatments but with slightly different intensities, it may be a good starting point to discuss with the patients their diabetes treatment, taking into account both the intensity of treatment, clinical factors and patients' preferences. The aim of the study was to evaluate whether such an approach increases the proportion of treatment goals that T2DM patients achieve.

Methods: In a cluster-randomised trial in 40 primary care practices that participated until 2009 in the ADDITION Study, 150 T2DM patients 60 - 80 years, known with T2DM for 8-15 years, will be included. Practices are randomised a second time, i.e. intervention practices in the ADDITION study could be control practices in the current study and vice versa. For the GPs from the intervention group a 2-hour training in shared decision making (SDM) was developed as well as a decision support tool to use during the consultation. These GPs plan the first visit with the patients to decide on the intensity of the treatment, personalised targets and the priorities of treatment. The control group will continue with the treatment they were allocated to in the ADDITION study (treatment-as-before). Follow-up: 24 months. The primary outcome is the proportion of patients who achieve all three treatment goals (HbA1c, blood pressure, total cholesterol) at 24 months. Secondary outcomes are the proportion of patients who achieve five treatment goals (HbA1c, blood pressure, total cholesterol , body weight, not smoking), evaluation of the SDM process (SDM-Q9), satisfaction with the treatment (DTSQ), wellbeing and quality of life (W-BQ12, ADD QoL-19), health status (SF-36, EQ-5D) and coping (DCMQ). The proportions of achieved treatment goals will be compared between groups by estimating the relative risk of meeting the treatment targets. For the secondary outcomes mixed models will be used.

Discussion: To achieve optimal diabetes care with a higher proportion of achieved individualised treatment goals, the SDM approach including a multi-faceted decision support tool might be useful. An intervention with such a support decision tool is designed.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Two more or less comparable categories of patients are eligible: 1. if diagnosed with T2DM in 2002-2004 by screening, aged between 50-70 years at that time and having participated in the ADDITION-study that ended in 2009; 2. treated for their T2DM in a practice that participated in the ADDITION study, between 60 and 80 years in 2012-2014 and with a T2DM duration between 8 to 15 years.

Exclusion Criteria:

* Patients will be excluded if they have a history of alcoholism, drug abuse, psychosis, personality disorder or another emotional, psychological or intellectual problem that is likely to invalidate informed consent, or limit the ability of the individual to comply with the protocol requirements and patients with a limited life expectancy.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The between groups difference in the proportion of patients which achieve the treatment goals for HbA1c, blood pressure, and total cholesterol | after 12 months
  The proportions of achieved treatment goals of HbA1c, blood pressure, total cholesterol within each study group will by estimated by calculating relative risk. Intention-to-treat analyses (ITT) will be performed to examine between-group differences.

SECONDARY OUTCOMES:
The difference between groups in the proportion of patients which achieved the five treatment goals for HbA1c, blood pressure, total cholesterol, body weight, and smoking. | after 24 months
  The proportions of achieved treatment goals of HbA1c, blood pressure, total cholesterol, body weight, and smoking, within each study group will by estimated by calculating relative risk.
Characteristics of success for the SDM process in the patients in the intervention group. | after 24 months
  Generalized linear models will be used to correct for clustering at practice level. To identify patients who show better results after the SDM process, the analysis for the primary outcome will be repeated with taking into account interaction of SDM with age, gender, education level, duration of diabetes.
The difference in health related Quality of Life between both groups at 24 months as measured with the Audit of Diabetes Dependent Quality of Life and the European Quality of Life questionnaire. | after 24 months
  The ADDQoL-19 measures the perceived impact of diabetes on the quality of life and includes 19 items. Items range from -3 to 3 on different questions, with 0 as the neutral score. Scores below 0 reflect a negative influence of the item on quality of life, and all above 0 reflect positive influences. The EQ-5D covers 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a Visual Analogue Scale (VAS) where respondents can rate their health. Item scores range from 1-3, and a 5-digit health profile is formed, placing the 5 numbers behind each other.
  Difference in health-related quality of life between baseline and 24 months follow-up within each group will be analysed by using paired t-tests. Mixed models will be used to study the between groups differences after two years. We will add random effects for patient and practice.
The difference in health status between both groups at 24 months as measured with the Short Form-36. | after 24 months
  The Short Form-36 (SF-36) is 36-item instrument for the self-evaluation of health status; it includes eight subscales: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. These scales can be summarised in Physical Health and Mental Health. The 36 items differ in the scoring ranges.
  Difference in health status between baseline and 24 months follow-up within each group will be analysed by using paired t-tests. Mixed models will be used to study the between groups differences after two years. We will add random effects for patient and practice.
The difference in well-being between baseline and 24 months within and between both groups as measured with the Well-Being Questionnaire. | after 24 months
  The Well-Being Questionnaire (W-BQ12) consists of 12-items in three 4-item subscales: negative well-being (item 1-4, higher score reflects a greater sense of negative well-being), energy (items 6 and 7 are reversed, and then together with 5 and 8 form the total amount of energy) and positive well-being (items 9-12, the higher the score the greater the sense of positive well-being). The total score ranges from 0 to 36 and is called the general well-being score. Higher scores indicate a higher overall sense of well-being.
  Difference in wellbeing between baseline and 24 months follow-up within each group will be analysed by using paired t-tests. Mixed models will be used to study the between groups differences after two years. We will add random effects for patient and practice.
The difference in wellbeing between baseline and 24 months within and between both groups as measured with the Well-Being Questionnaire. | after 24 months
  The Well-Being Questionnaire (W-BQ12) consists of 12-items in three 4-item subscales: negative well-being (item 1-4, higher score reflects a greater sense of negative well-being), energy (items 6 and 7 are reversed, and then together with 5 and 8 form the total amount of energy) and positive well-being (items 9-12, the higher the score the greater the sense of positive well-being). The total score ranges from 0 to 36 and is called the general well-being score. Higher scores indicate a higher overall sense of well-being.
  Difference in wellbeing between baseline and 24 months follow-up within each group will be analysed by using paired t-tests. Mixed models will be used to study the between groups differences after two years. We will add random effects for patient and practice.
The difference in coping style between baseline and 24 months within and between both groups as measured with the Diabetes Coping Measurement Questionnaire. | after 24 months
  The Diabetes Coping Measurement Questionnaire (DCMQ) consists of 21 items. Overall scores range from 7 to 35. The items are measures on a 5-point Likert scale, ranging from 1 ("disagree") to 5 ("agree strongly") or from 1 ('I strongly agree') to 5 (I 'disagree'). It includes 4 subscales: spirit coping, avoidance coping, passive resignation coping and diabetes integration coping. Higher scores on tackling spirit and diabetes integration indicate more adaptive coping. Higher scores on passive resignation and avoidance indicate poor coping.
  Difference in coping style between baseline and 24 months follow-up within each group will be analysed by using paired t-tests. Mixed models will be used to study the between groups differences after two years. We will add random effects for patient and practice.

OTHER OUTCOMES:
Process evaluation of the shared decision making ability of the general practitioners by using the Shared Decision Making Questionnaire. | at 24 months
  The Shared Decision Making Questionnaire (SDM-Q9) includes 9 items with ratings from 0 (completely disagree) to 6 (completely agree); the total score ranges from 0 to 45.
  The shared decision making ability of the general practitioners in both the intervention and the control practices (the first group trained, the latter not trained) will be evaluated during the final measurement occasion (24 months) by using the SDM-Q9, filled out by both the patients and the general practitioners. In addition, one or two audio tabs per GP including a selection of the SDM visit will be analysed, as well as some of the final visits in the control practices. These audio tabs will be evaluated by two independent observers by using the SDM-Q9.

CONTACTS AND LOCATIONS:
Overall Officials: Guy EH Rutten, MD PhD, Principal Investigator — Julius Centre
Locations (1):
- Julius Centre for Health Sciences and Primary Care, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
no plan yet, but for data request the authors can be contacted

REFERENCES:
- [Background] Griffin SJ, Borch-Johnsen K, Davies MJ, Khunti K, Rutten GE, Sandbaek A, Sharp SJ, Simmons RK, van den Donk M, Wareham NJ, Lauritzen T. Effect of early intensive multifactorial therapy on 5-year cardiovascular outcomes in individuals with type 2 diabetes detected by screening (ADDITION-Europe): a cluster-randomised trial. Lancet. 2011 Jul 9;378(9786):156-67. doi: 10.1016/S0140-6736(11)60698-3. Epub 2011 Jun 24. PMID 21705063
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Background] Stiggelbout AM, Van der Weijden T, De Wit MP, Frosch D, Legare F, Montori VM, Trevena L, Elwyn G. Shared decision making: really putting patients at the centre of healthcare. BMJ. 2012 Jan 27;344:e256. doi: 10.1136/bmj.e256. PMID 22286508
- [Background] Wilkinson MJ, Nathan AG, Huang ES. Personalized decision support in type 2 diabetes mellitus: current evidence and future directions. Curr Diab Rep. 2013 Apr;13(2):205-12. doi: 10.1007/s11892-012-0348-6. PMID 23160795
- [Derived] den Ouden H, Vos RC, Reidsma C, Rutten GE. Shared decision making in type 2 diabetes with a support decision tool that takes into account clinical factors, the intensity of treatment and patient preferences: design of a cluster randomised (OPTIMAL) trial. BMC Fam Pract. 2015 Feb 27;16:27. doi: 10.1186/s12875-015-0230-0. PMID 25887759